CLINICAL TRIAL: NCT04774523
Title: Evaluation of the BIOTRONIK AutoAdapt Algorithm for Continuous Automatic Adaptive Cardiac Resynchronization
Acronym: BIO|Adapt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR028
Record Dates: First submitted 2021-02-19; First posted 2021-03-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Cardiac Arrhythmia; Left Ventricular Dysfunction
Keywords: CRT therapy; Heart Failure; AV optimization; Left Ventricular Ejection Fraction; AutoAdapt algorithm
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: There will be two arms with the same study flow chart along the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): This group will be made up of patients implanted with CRT-D devices without the CRT AutoAdapt feature, or with the CRT AutoAdapt feature deactivated.
  Interventions: Procedure: Echocardiography AV optimization; Procedure: Echocardiography; Other: Self Assessment Score
- AutoAdapt group (Experimental): This group will be made up of patients implanted with CRT-D devices that have the CRT AutoAdapt feature available. It is mandatory that all patients within this group have the feature activated, independently of other characteristics.
  Interventions: Procedure: Echo-based assessment of the acute hemodynamic effect of the CRT AutoAdapt feature.; Procedure: Echocardiography; Other: Self Assessment Score

INTERVENTIONS:
Procedure: Echo-based assessment of the acute hemodynamic effect of the CRT AutoAdapt feature. — Patients in the AutoAdapt group undergo the echo-based assessment of the acute hemodynamic effect of the CRT AutoAdapt feature.
  Three steps must be followed:
  1. Standard AV programming: perform echo for AoVTI assessment.
  2. Echo-optimized AV programming: perform standard echo-based AV-optimization (Ritter method or iterative method, according to routine at investigational site); measure AoVTI at optimized setting.
  3. AutoAdapt optimized programming: The system allows different programming options for the parameter 'Adaptive AV reduction'. The nominal value is 0.7, but it can be modified to different values ranging from 0.5 to 0.9. The AoVTI shall be measured at standard setting of the "Adaptive Av reduction" parameter, 0.7.
  Arms: AutoAdapt group
Procedure: Echocardiography AV optimization — Patient in the control group undergo the routine echo-based AV-optimization that is usually performed at the investigational site (Ritter method or iterative method). Performance of an additional VV-delay optimization is left to the investigator discretion
  Arms: Control group
Procedure: Echocardiography — Echocardiography must be performed at baseline and 12 month Follow Up to collect the LVEF/LVESD(V)/LVEDD(V)
Other: Self Assessment Score — Patient must complete the self assessment score at 6 and 12 month Follow Up, that will be use for the Packer Clinical Composite Score

SUMMARY:
BIO|Adapt study is designed to provide evidence for the clinical benefit of the CRT AutoAdapt feature. This feature provides continuous adaptation of AV delay and biventricular pacing modality. However, additional clinical data on the short and mid-term improvement of CRT-D patients by the CRT AutoAdapt feature are needed.

DETAILED DESCRIPTION:
The magnitude of clinical and hemodynamic benefit of CRT varies significantly among its recipients. Many studies report that approximately one-third of the implanted population show no clinical improvement at follow-ups. There are many clinical factors that are associated with the CRT response and the grade of benefit, such as type of cardiomyopathy, severity of electrical conduction abnormalities, dyssynchrony, and scar burden. In addition, there are device-related factors such as lead location, insufficient ventricular pacing percentage (%V), and suboptimal atrial-ventricular (AV) and ventricle- ventricle (VV) timing.

The main finding in such CRT non-responders is a suboptimal AV-timing (47%). The optimization of AV and VV intervals during biventricular (BiV) pacing is an option to maximize the positive effects of CRT, by taking advantage of the full atrial contraction for optimal filling of the ventricles. Optimization is usually accomplished by using echocardiography or other methods. However, such methods are time consuming for the hospitals and may not provide a benefit for every patient.

The most common pacing mode for CRT therapy is BiV pacing, but many acute and chronic randomized clinical studies have demonstrated that left-ventricular (LV) pacing can be at least as effective as BiV pacing. In patients with sinus rhythm and normal atrioventricular (AV) conduction, pacing the left ventricle only with an appropriate AV interval can result in an even superior LV and right ventricular (RV) function compared with standard BiV pacing. LV pacing has been proposed as an alternative approach to apply cardiac resynchronization as it has been shown that LV pacing induces short-term hemodynamic benefits compared to BiV pacing.

Different algorithms have been developed by different manufactures to provide continuous automatic CRT optimization, allowing a more physiologic ventricular activation and greater device longevity in patients with normal AV conduction due to the reduction of unnecessary RV pacing. Studies with the Medtronic Adaptive cardiac resynchronization therapy (aCRT) algorithm, that provides automatic ambulatory selection between synchronized LV or BiV pacing with dynamic optimization of atrioventricular and interventricular delays, have shown that the algorithm is safe and as effective as BiV pacing with comprehensive echocardiographic optimization.

The CRT AutoAdapt feature by BIOTRONIK optimizes the CRT therapy settings of the device automatically and continuously. This algorithm adjusts the AV delay and sets the ventricular pacing configuration to BiV or LV. The settings are based on intracardiac conduction times, which are measured every 60 seconds to select the optimal configuration.

The objective of this study is to show non-inferiority of this feature compared to standard echo-based optimization with regard to clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Indication for de novo implantation or upgrade to a CRT-D device
* Enrolled in BIO|STREAM.HF but not yet implanted with or upgraded to CRT-D
* LVEF < 35%
* QRS > 120 ms
* NYHA II-IV
* Atrial heart rate during sinus rhythm at rest below 100 bpm
* Patient is able to understand the nature of the study and willing to provide written informed consent to this submodule

Exclusion Criteria:

* Planned implantation or previous implantation with a BIOTRONIK DX ICD lead
* History of persistent/permanent AF
* History of complete AV-block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
CRT-responder rate based on improvement in Clinical Composite Score developed by Packer at 12 month follow up. | 12 month Follow Up
  It will be use Packer Score to assess the clinical outcome in heart failure patients. It takes into account all possible dimensions of outcome, i.e. mortality, morbidity and quality of life and is based on the following data points:
  * Death (yes/no)
  * Any unplanned hospitalization for worsening heart failure (yes/no)
  * Change in NYHA class compared to baseline (improved/unchanged/worsened)
  * Patient's global assessment (PGA) compared to baseline (improved - three stages / unchanged / worsened - three stages)
  * Discontinuation of study protocol due to worsening heart failure, treatment failure or lacking therapeutic response (yes/no)
  At the end of the study, the outcome of each patient is classified as:
  * Worsened
  * Unchanged
  * Improved

SECONDARY OUTCOMES:
Acute hemodynamic effect of AutoAdapt feature | At pre-hospital discharge assessed up to 30 days since the implantation
  The acute hemodynamic response to different parameter settings will be assessed by measuring the aortic velocity time integral (AoVTI) via echocardiography.
Change in LVEF | 12 month Follow Up
  The intra-individual change in LVEF from baseline to 12 month FU will be assessed by echocardiography as a measure of improvement in cardiac function and compared between patient groups.
Change in Left Ventricular End Diastolic and Systolic Diameter (LVED(S)D) | 12 month Follow Up
  The intra-individual change in LVED(S)D from baseline to 12 month FU will be assessed by echocardiography as a measure of ventricular reverse remodeling and compared between patient groups.
Change in Left Ventricular End Diastolic and Systolic Volumes (LVED(S)V) | 12 month Follow Up
  The intra-individual change in LVED(S)V from baseline to 12 month FU will be assessed by echocardiography as a measure of ventricular reverse remodeling and compared between patient groups.
Change in NYHA class | 12 month Follow Up
  The intra-individual change in the NYHA classification from baseline to 12 months will be assessed as a measure of overall functional improvement and compared between patient groups.
Percentage of LV only pacing | 12 month Follow Up
  The percentage of LV only pacing based on device statistics will be assessed at the 12 months FU and compared between patient groups to assess the potential to reduce battery consumption by the AutoAdapt feature.
Adverse device effects related to the CRT AutoAdapt feature | 12 month Follow Up
  Evaluation of all reported adverse device effects for a possible relation with the CRT AutoAdapt feature

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier García Fernandez, Physician, Principal Investigator — Hospital Universitario de Burgos, Spain
Locations (1):
- Dr Francisco Javier Garcia, Burgos, Castille and León, Spain